CLINICAL TRIAL: NCT06826391
Title: Evaluating the Use of Calcium Hydroxylapatite With Integral Lidocaine for Improving Gingival Recession and Hypersensitivity
Brief Title: Using Calcium Hydroxylapatite To Treat Gum Recession and Tooth Hypersensitivity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Facial Esthetics (Network)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2025-02-09; First posted 2025-02-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Gingival Recession, Generalized; Gingival Recession Generalized Moderate; Gingival Recession Localized Moderate; Tooth Sensitivity
Keywords: Gingival recession; Tooth sensitivity; Recessed gums; Gum recession; Attached gingiva; Attached gingiva deficiency
MeSH Terms: conditions — Gingival Recession; Dentin Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Evaluating the Use of Calcium Hydroxylapatite For Improving Gingival Recession and Hypersensitivity (Experimental): * The dentist determines the tooth/teeth to be treated, the patient will receive injections of a numbing agent to numb the gums.
  * Once the patient is numb, he/she will be injected with Radiesse+ on each affected tooth/teeth and one additional tooth on each side of affected tooth/teeth in approximately 5 injection sites per affected tooth in the following locations: papilla (gum between two teeth), halfway between papilla and apex, apex, halfway between papilla on the other side of the tooth and apex, and the second papilla.
  Interventions: Device: Calcium hydroxylapatite

INTERVENTIONS:
Device: Calcium hydroxylapatite — This intervention consists of calcium hydroxylapatite injections into the attached gingiva of a patient who has gingival recession to stabilize, grow and reverse gingival recession. These injections will also reduce tooth hypersensitivty in the affected teeth.

SUMMARY:
Study Purpose and Objectives:

This study will utilize calcium hydroxylapatite (CaHA) to treat recession and hypersensitivity of the gums.

The objectives of the study are:

1. to study the quality and quantity of changes in attached gums resulting from Radiesse(+) injections in the gingival tissue;
2. to determine the efficacy of Radiesse(+) in the reduction of tooth hypersensitivy caused by exposed roots relating to gingival recession;
3. to determine the efficacy of Radiesse(+) in the treatment of mild and moderate gingival recession.

DETAILED DESCRIPTION:
Recession of the gingiva or gums, is a prevalent condition in the U.S. population. Gum recession can start early in life, with ~27% of people 15-25 years experiencing recession. The frequency of gum recession increases with age, with 70.3% of adults 45-60 years and ~100% of adults will experience gum recession in their lifetime.

Recession of the gums is defined as the shift of the marginal gingiva from its normal position on the crown of the tooth to the levels on the root surface beyond the cemento-enamel junction.

Whereas many dental conditions go unnoticed by patients, gum recession can often be visible to patients and for which they may seek advice of a dentist. Gingival recession of the front teeth usually creates an aesthetic problem and anxiety about tooth loss due to progression of the destruction.

Gum recession may also be associated with dentin hypersensitivity, root caries, abrasion and/or cervical wear, erosion because of exposure of the root surface to the oral environment and an increase in accumulation of dental plaque.

Gum recession may be caused by a variety of factors, including but not limited to smoking, hormonal changes, genetics, periodontal disease or insufficient dental hygiene. Treatment for gum recession includes a deep cleaning, dental bonding, antibiotics and surgery.

Calcium hydroxylappetite (CaHA; Radiesse, Merz Aesthetics, Raleigh, NC) is FDA cleared as a facial implant for volume improvement for moderate to severe wrinkles and folds such as the nasolabial folds. CaHA is also cleared by the FDA to fill and/or augment dental defects, including periodontal defects.

Radiesse is composed of synthetically produced, smooth and uniform calcium hydroxide microspheres suspended in carboxymethylcellulose gel in ratio 30% microspheres to 70% gel by volume. Radiesse(+) and is the same formulation as Radiesse with the addition of lidocaine in powder format, which reduces pain of injection.

The CaHA in Radiesse/Radiesse(+) is biocompatible and possess a low risk of stimulating an immune response. Studies have shown that CaHA is an effective collagen and elastin stimulator as well as a robust filler for soft tissue augmentation. CaHA has recently been shown to improve gum recession with results that lasted 6 months and up to 12 months6, as well as resulted in a reduction in gum hypersensivity.

ELIGIBILITY:
Inclusion Criteria:

* • Patient selection criteria will be limited to male or female patients between the ages of 20-70 years old.

  * Patient must be in good medical health
  * Patient has no active periodontal gum disease or inflammation of the gums
  * Has thin or intermediate gum collar around the teeth
  * Has mild to moderate gum recession as determined by the AAFE Gingival Recession Classification
  * Tooth/teeth to be treated for this study to include teeth numbers 5 - 12 and 21 - 28 (see image below)
  * Written informed consent has been obtained
  * Written authorization for Use and Release of Health and Research Study Information has been obtained
  * Ability to follow study instructions and likely to complete all required visits
  * If the subject is female of childbearing potential (sexually active and not sterile, surgically sterilized, or postmenopausal with no menses for a least 1 year), the subject has used contraception for at least 30 days prior to enrollment and agrees to use a reliable method of contraception (birth control pills, has an intrauterine device (IUD), and/or condoms) for the duration of the study.

Exclusion Criteria:

* • Uncontrolled systemic disease

  * Known allergy or sensitivity to the study medication or its components
  * Females who are pregnant, nursing, or planning a pregnancy
  * Current enrollment in another investigational drug or device study or participation in such a study within 30 days of entry into this study and for the duration of the study
  * Infection at the injection sites
  * Evidence of recent alcohol or drug abuse
  * Has a history of severe allergic reactions or allergy to numbing agents
  * Has an active inflammation, infection, cancerous or precancerous lesion, or unhealed wound in the mouth
  * History of trauma associated with the teeth and/or mouth that in the judgment of the investigator may affect evaluation of safety or efficacy of treatment
  * Presence of any clinically significant bleeding disorder or is receiving medication that will likely increase the risk of bleeding as the result of injection (subjects being treated with antiplatelet therapy, anticoagulants and acetylsalicylic acid could be enrolled after 7-day washout period
  * Subject has a condition or is in a situation which, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
  * Any medical condition (e.g., respiratory, cardiovascular, hepatic, neurological disease, or thyroid dysfunction) or psychiatric disorders (including schizophrenia, bipolar, major depressive, obsessive compulsive, post traumatic stress, borderline personality, panic) that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Of Gingival Recession With Calcium Hydroxylapatite Injections In Attached Gingiva | 3 months
  Gum recession will be measured at baseline, during the study, and at the end of the study for the affected teeth. For gum recession, a dentist will measure the amount of gum recession present at each stage. Gum recession measurements range from 0 -10 mm. 0 means no gum recession and 10 is severe gum recession.
  Investigators and patients will grade their results based on the Global Aesthetic Improvement Scale (GAIS) as (1) very much improved, (2) much improved, (3) improved, (4) no change. The same doctor will be taking the measurements and administering treatment at each stage to standardize the information in this study.
Change from Baseline Of Tooth Hypersensitivity With Calcium Hydroxylapatite Injections In Attached Gingiva | 3 months
  Tooth hypersensitivity will be measured at baseline, during the study, and at the end of the study for the affected teeth. Tooth hypersensitivity will be assessed by the patient on a 0-10 scale at each stage of the study. Zero is equivalent to no pain and 10 indicates the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Louis Malcmacher, DMD, Principal Investigator — American Academy of Facial Esthetics
Locations (1):
- American Academy of Facial Esthetics, South Euclid, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Specific individual participant data sets to be shared will include the study protocol, the statisical analysis plan, the informed consent form, adverse reaction form, the clinical study report, analytic codes if any, all collected IPD, and all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The time frame will be beginning 3 months and ending 3 years after the publication of results
Access Criteria: The criteria that will be met in order for data to be shared includes statistical methods which must be approved by independent review. A proposal that describes planned analyses must be submitted. A data sharing agreement must be signed. These documents can be submitted to the Primary Investigator, Dr. Louis Malcmacher, who will review requests for IPD sharing.

REFERENCES:
- [Background] Roccuzzo M, Bunino M, Needleman I, Sanz M. Periodontal plastic surgery for treatment of localized gingival recessions: a systematic review. J Clin Periodontol. 2002;29 Suppl 3:178-94; discussion 195-6. doi: 10.1034/j.1600-051x.29.s3.11.x. PMID 12787218
- [Background] Nieri M, Pini Prato GP, Giani M, Magnani N, Pagliaro U, Rotundo R. Patient perceptions of buccal gingival recessions and requests for treatment. J Clin Periodontol. 2013 Jul;40(7):707-12. doi: 10.1111/jcpe.12114. Epub 2013 May 13. PMID 23668251
- [Background] Renkema AM, Fudalej PS, Renkema A, Bronkhorst E, Katsaros C. Gingival recessions and the change of inclination of mandibular incisors during orthodontic treatment. Eur J Orthod. 2013 Apr;35(2):249-55. doi: 10.1093/ejo/cjs045. Epub 2012 Jul 24. PMID 22828081
- [Background] Agudio G, Nieri M, Rotundo R, Franceschi D, Cortellini P, Pini Prato GP. Periodontal conditions of sites treated with gingival-augmentation surgery compared to untreated contralateral homologous sites: a 10- to 27-year long-term study. J Periodontol. 2009 Sep;80(9):1399-405. doi: 10.1902/jop.2009.090122. PMID 19722789
- [Background] Kennedy JE, Bird WC, Palcanis KG, Dorfman HS. A longitudinal evaluation of varying widths of attached gingiva. J Clin Periodontol. 1985 Sep;12(8):667-75. doi: 10.1111/j.1600-051x.1985.tb00938.x. PMID 3902907
- [Background] Shalak OV, Satygo EA. The effectiveness of calcium hydroxylapatite-based implant in eliminating increased sensitivity of teeth. Herald of North-Western State Medical University named after I.I. Mechnikov. 2024;16(1):79-86
- [Background] Shalak OV, Satygo EA, Deev RV, Presnyakov EV. The efficacy of Radiesse(+) in dental practice for prevention and non-surgical treatment of gingival recession. Herald of North-Western State Medical University named after I.I. Mechnikov. 2022;14(4):43-52.
- [Background] 5. Shawky HA, Darwish MM. Clinical application of Radiesse(+) and hyaluronic acid gel for treatment of papillae deficiencies in the esthetic zone. Egyptian Dental J. 2017;63:533-545.
- [Background] Loe H, Anerud A, Boysen H. The natural history of periodontal disease in man: prevalence, severity, and extent of gingival recession. J Periodontol. 1992 Jun;63(6):489-95. doi: 10.1902/jop.1992.63.6.489. PMID 1625148
- [Background] Mythri S, Arunkumar SM, Hegde S, Rajesh SK, Munaz M, Ashwin D. Etiology and occurrence of gingival recession - An epidemiological study. J Indian Soc Periodontol. 2015 Nov-Dec;19(6):671-5. doi: 10.4103/0972-124X.156881. PMID 26941519
- See also: Causes and treatments for gum recession — https://www.webmd.com/oral-health/receding_gums_causes-treatments